CLINICAL TRIAL: NCT07370337
Title: Phase II, Single-Arm, Multicenter Clinical Study of Induction Chemotherapy Combined With Tislelizumab as Neoadjuvant Therapy for Locally Advanced Squamous Cell Carcinoma of the External Auditory Canal
Brief Title: Induction Chemotherapy Combined With Tislelizumab for Locally Advanced Squamous Cell Carcinoma of the External Auditory Canal
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xinmao Song, Associate chief physician, Eye & ENT Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025029
Record Dates: First submitted 2026-01-13; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma of External Auditory Canal; Locally Advanced Tumor
MeSH Terms: interventions — tislelizumab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction Chemotherapy Combined with Tislelizumab for Locally Advanced SCC of the EAC (Experimental)
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Eligible patients will receive 2-3 cycles of neoadjuvant therapy consisting of tislelizumab combined with the AP chemotherapy regimen (nab-paclitaxel+ cisplatin).
  Other Names: Neoadjuvant chemotherapy

SUMMARY:
To evaluate the efficacy and safety of induction chemotherapy combined with tislelizumab as neoadjuvant therapy in patients with locally advanced squamous cell carcinoma of the external auditory canal; to explore the improvement in the preservation rate of important neurovascular structures (including the facial nerve, internal carotid artery canal, sigmoid sinus, and posterior cranial nerves, etc.).

DETAILED DESCRIPTION:
The main reasons for the poor prognosis of advanced squamous cell carcinoma of the external auditory canal are the strong local invasiveness of the tumor, the complexity of the adjacent anatomical structures, the high difficulty in complete tumor resection, and the imperfection of comprehensive treatment strategies. In this phase II single-arm clinical study, the investigators aimed to evaluate the efficacy and safety of induction chemotherapy (nab-paclitaxel plus cisplatin) combined with tislelizumab as neoadjuvant therapy in patients with locally advanced squamous cell carcinoma of the external auditory canal, and to explore the improvement in the preservation rate of important neurovascular structures (including the facial nerve, internal carotid artery canal, sigmoid sinus, posterior cranial nerves, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old and ≤ 80 years old
2. Pathologically confirmed as squamous cell carcinoma
3. Suitable for enhanced MRI/CT imaging assessment
4. Previously untreated squamous cell carcinoma of the external auditory canal staged as cT3-4NxM0 according to the Pittsburgh clinical staging system
5. Cases that meet the inclusion criteria following joint discussion with otologists
6. Expected survival time of at least 1 year
7. ECOG performance status score of 0-1
8. Peripheral blood routine examination before treatment meets the following criteria: neutrophil count > 2,000/mm³; platelet count > 100,000/mm³
9. Liver and kidney function tests before treatment meet the following criteria: bilirubin < 1.5 mg/dl; AST or ALT < 1.5 × upper limit of normal (ULN); serum creatinine < 1.5 mg/dl; creatinine clearance rate > 60 ml/min
10. Signed informed consent form prior to the initiation of the study

Exclusion Criteria:

1. Ear tumors whose pathological type is not squamous cell carcinoma
2. Patients with early-stage (T1-T2) disease or distant metastasis (M1)
3. Cases not jointly discussed with an otologist
4. Non-first-time radiotherapy for the head and neck region
5. Hypersensitivity to platinum-based drugs or taxane drugs
6. A history of head and neck malignant tumors, or concurrent multiple primary tumors
7. Positive pregnancy test result in women of childbearing age
8. Concurrent diseases or conditions that affect the patient's normal enrollment or safety during the study period
9. Active mental disorders or other psychological conditions that impair the patient's ability to sign the informed consent form and comprehend study-related information
10. Uncontrolled active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | Two weeks after Induction Therapy
  Objective Response Rate after Induction Therapy
Preservation Rate of Neurovascular Function | Immediately after surgery
  Preservation Rate of Neurovascular Function (Facial Nerve, Carotid Artery Canal, Sigmoid Sinus, Posterior Cranial Nerves)

SECONDARY OUTCOMES:
Disease-free survival ( DFS) | 2 year
Overall survival （OS） | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Li Wang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided